CLINICAL TRIAL: NCT04463238
Title: Randomized Open Multicenter Clinical Study to Evaluate the Safety and Effectiveness of Guided Cartilage Regeneration Membrane for Repair of Articular Cartilage Injury
Brief Title: Guided Cartilage Regeneration Membrane
Acronym: GCRM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Zhongnan Hospital (Other); Second Hospital of Shanxi Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); First Affiliated Hospital of Kunming Medical University (Other); Zunyi Medical College (Other); The First Affiliated Hospital of Zhengzhou University (Other); Chinese PLA General Hospital (Other); Xi'an Honghui Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015035
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Articular Cartilage Injury; Knee Ligament Injury
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Intervention Model Description: GCRM-3020\GCRM-4030
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cartilage membrane surgery (Experimental): The test group applied the guidance provided by Shaanxi Baiao Regenerative Medicine Co., Ltd.
  Cartilage regeneration membrane combined with microfracture surgery.
  Interventions: Combination Product: Guided cartilage regeneration membrane; Procedure: Microfracture
- Microfracture (Other): The control group was treated with microfractures widely recognized at home and abroad.
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Combination Product: Guided cartilage regeneration membrane — On the basis of microfracture, the blood clot released from the defect area is covered with a guide cartilage regeneration membrane to provide an attached scaffold for the cells in the blood clot.
  Arms: Cartilage membrane surgery
Procedure: Microfracture — Operate in accordance with the clinical microfracture surgery method.

SUMMARY:
Guided cartilage regeneration membrane for repairing the safety and effectiveness of articular cartilage injury

DETAILED DESCRIPTION:
MRI evaluation using guided cartilage regeneration membrane for articular cartilage injury repair 730 days (2 years) is the main indicator of this trial. In this experiment, we observe the improvement of Lysholm score, VAS score, ratio change of regenerated cartilage T2 value to normal cartilage T2 value, and ratio of regenerated cartilage △R1 value to normal cartilage △R1 value Indicators such as value changes are secondary evaluation indicators.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old and ≤50 years old, regardless of gender
2. 2 cm2 ≤ articular cartilage defect repair area ≤ 8 cm2, patients with feasible micro-fractures, no contraindications to surgery
3. Patients voluntarily participate in clinical trials, sign informed consent forms, and can cooperate with clinical follow-up

Exclusion Criteria:

1. Those who have participated in clinical trials of other drugs or medical devices in the last 6 months
2. Those with stage III or above degeneration of bone and joint
3. Those who cannot accept pig-derived devices or have special religious beliefs due to religion, ethnicity and other issues
4. Those who are sensitive to collagen, foreign protein or pig-derived materials
5. Repair the damaged area> 8 cm2 or <2 cm2, lack of normal cartilage tissue around the injury
6. Severe heart, liver and kidney insufficiency are defined as:

   Heart function: NYHA grade III or above; ALT, AST> 2.5 times the upper limit of normal value; Serum creatinine> 1.5 times the upper limit of normal value;
7. People with systemic immune diseases or systemic or local infections
8. Joint fibrosis, joint stiffness, and obviously restricted movement
9. Those with moderate or severe osteoarthritis
10. People with contraindications for MRI examination
11. Patients with hemophilia
12. Those who cannot tolerate surgery
13. Women who are pregnant or plan to become pregnant and breastfeeding women
14. Persons with mental abnormalities and incapacity to act autonomously
15. Other conditions that the doctor judges cannot participate in the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-03 (Estimated); Primary Completion 2022-08-03 (Estimated); Study Completion 2023-08-03 (Estimated)

PRIMARY OUTCOMES:
MRI evaluation of articular cartilage injury 730 days (2 years) after repair | End of surgery to 730 days after surgery
  The nuclear magnetic evaluation indicators are as follows:
  1. Cartilage defect repair filling degree;
  2. Fusion of repair tissue and adjacent normal cartilage;
  3. Repair tissue surface structure;
  4. Repair the internal structure of the organization.
  The MRI score of the experimental group before and after treatment increased by an average of 5 points compared with the control group.

SECONDARY OUTCOMES:
Change in ratio of regenerated cartilage T2 value to normal cartilage T2 value | At 24 months after surgery
  The closer the ratio of the regenerated cartilage T2 value to the normal control cartilage T2 value is 1, it means that the regenerated cartilage The closer the water content and collagen arrangement are to normal cartilage.
Change in ratio of regenerated cartilage △R1 value to normal cartilage △R1 value | At 24 months after surgery
  The closer the ratio of the regenerated cartilage △R1 value to the normal control cartilage △R1 value is 1, it means that the GAG content of regenerated cartilage is closer to normal cartilage.

CONTACTS AND LOCATIONS:
Overall Officials: Yingfang Ao, PhD, Principal Investigator — Department of Sports Medicine, Peking University Third Hospital; Xiaoqing Hu, PhD, Study Director — Department of Sports Medicine, Peking University Third Hospital
Locations (8):
- China (8):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Zunyi Medical College, Zunyi, Guizhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongnan Hospital, Wuhan, Hubei
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xi'an Honghui Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Kunming Medical College, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No